CLINICAL TRIAL: NCT01188161
Title: The Effects of Whole Body Rotations in the Pitch and Yaw Planes on Postural Stability
Brief Title: Postural Effects of Being Rotated in a Whole Body Gyroscope
Acronym: Gyro
Status: Completed | Type: Observational
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Prof Frederick Carrick, Carrick Institute for Graduate Studies
Other Study IDs: 1-2010-06
Record Dates: First submitted 2010-08-20; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Falls; Balance; Movement Disorders
Keywords: Posturography; Balance; Falls; Gyroscope; Rotational Chair; Vestibular; Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normal subjects: Volunteers without a history of dizzyness or vertigo
  Interventions: Device: Rotating Chair

INTERVENTIONS:
Device: Rotating Chair — Subjects will be spun in rotating chair
  Other Names: gyrostim

SUMMARY:
Subjects will be secured and rotated in a whole body gyroscope, similar to a flight trainer for astronauts. The rotations will be in many directions and the speed will be at 90 deg/sec. The effects of this rotation on the ability to stand upright will be measured.

DETAILED DESCRIPTION:
Computerized dynamic posturography (CDP) testing will be obtained after practice sessions on all subjects using a CAPS Pro system (Vestibular Technologies, Cheyenne WY, USA). All tests will be conducted with the subject standing on a perturbing foam cushion. Six different conditions will be tested in sequence without the subjects stepping away from the foam/platform in order to assess if the center of sway position changed with the changing test conditions: (1) Eyes Open Head Neutral, (2) Eyes Closed Head Neutral, (3) Eyes Closed Head Right, (4) Eyes Closed Head Left, (5) Eyes Closed Head Flexed, (6) Eyes Closed Head Extended. Subjects will be continuously rotated in a computer-controlled multi-axis chair (Gyrostim by UltraThera Technologies, Inc.) in combinations of whole body Pitch and Yaw simultaneously over a 40 second profile at 90 deg/sec (15 RPM). The acceleration rates to 90 degrees per second as well as deceleration rates will be linear and occur in 1 second. We will utilize rotations that will represent all combinations of pitch and yaw with Pitch direction changing two times and Yaw direction four times (Backward Pitch -20 seconds with right Yaw-10 seconds to left Yaw-10 seconds, to Forward Pitch- 20 seconds with right Yaw-10 seconds to left Yaw 10 seconds). Post rotational CDP testing will be compared to the Pre Rotational CDP,

ELIGIBILITY:
Inclusion Criteria:

* Normal Healthy Adults without a history of vertigo or dizziness

Exclusion Criteria:

* History of dizziness or vertigo

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal healthy volunteers without a history of vertigo or dizziness
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Computerized Dynamic Posturography | 10 minutes after Rotation
  Standard platform posturography

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, Study Chair — Life University
Locations (1):
- Life University, Marietta, Georgia, United States